CLINICAL TRIAL: NCT01261663
Title: Impact of the Time of Oral Nutritional Supplements (ONS) Consumption on Daily Alimentary Intakes of Malnourished Elderly Subjects Hospitalized in Long Term Care Unit (LTCU)
Brief Title: Impact of the Time of Oral Nutritional Supplements (ONS) Consumption on Daily Alimentary Intakes of Malnourished Elderly
Acronym: ACTICLAN
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I09017
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Malnutrition in the Elderly

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NOS intake either at end of meals or as snackings.
  Interventions: Other: oral nutritional energy and protein enriched supplement (NOS)

INTERVENTIONS:
Other: oral nutritional energy and protein enriched supplement (NOS)

SUMMARY:
Malnutrition is a severe comorbidity in hospitalised patients, especially in elderly. The consumption of Oral Nutritional Supplements (NOS) is one of several tools for fighting against malnutrition. Their use is easy, and framed by recent French recommendations suggesting to propose NOS at end of meals or as snacking . Nevertheless, there is no scientific data to affirm which is the best of these two hypothesis in elderly hospitalised in Long Term Care Unit(LTCU) . Moreover, a preliminary survey of NOS consumption in LTCU in Limoges university hospital showed some problems about the mode of supplying NOS, partially linked with an insufficiency for paramedical staff in realizing importance of NOS. However, the effect of time of supplying NOS on total food consumption had not been evaluated in this first study. The new one will include 48 malnourished elderly patients in two LTCU and having a prescription of NOS. They will receive them at the same quantity during the whole study either firstly at end of meals (10 days) and secondly as snackings (10 days), or conversely. Order of choice will be randomised. Total daily alimentary intakes will be noted by paramedical staff of the two units, and translated by dieticians in daily energy, protein, carbohydrates and lipids intakes. The time of supplying NOS will be confronted with these intakes, in order to precise the best one.

DETAILED DESCRIPTION:
Malnutrition is a severe comorbidity in hospitalised patients, especially in elderly. The consumption of Oral Nutritional Supplements (NOS) is one of several tools for fighting against malnutrition. Their use is easy, and framed by recent French recommendations suggesting to propose NOS at end of meals or as snacking . Nevertheless, there is no scientific data to affirm which is the best of these two hypothesis in elderly hospitalised in Long Term Care Unit(LTCU) . Moreover, a preliminary survey of NOS consumption in LTCU in Limoges university hospital showed some problems about the mode of supplying NOS, partially linked with an insufficiency for paramedical staff in realizing importance of NOS. However, the effect of time of supplying NOS on total food consumption had not been evaluated in this first study. The new one will include 48 malnourished elderly patients in two LTCU and having a prescription of NOS. They will receive them at the same quantity during the whole study either firstly at end of meals (10 days) and secondly as snackings (10 days), or conversely. Order of choice will be randomised. Total daily alimentary intakes will be noted by paramedical staff of the two units, and translated by dieticians in daily energy, protein, carbohydrates and lipids intakes. The time of supplying NOS will be confronted with these intakes, in order to precise the best one.

ELIGIBILITY:
Inclusion Criteria:

* Malnourished elderly (age >=70 y) hospitalised in LTCU
* having a NOS medical prescription o

Exclusion Criteria:

* Non malnourished patients in LTCU,
* age <70.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Malnourished elderly (age >=70 y) hospitalised in long term care unit (LTCU)having a NOS medical prescription
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2014-06

PRIMARY OUTCOMES:
Total daily alimentary intakes | daily, for 20 consecutive days

SECONDARY OUTCOMES:
Protein, carbohydrates and lipids intakes | daily, for 20 consecutive days

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de Nutrition - Service hépato-gastro-entérologie, Limoges, France